CLINICAL TRIAL: NCT07313020
Title: A Visualization Clinical Study Using a Handheld MPI Imaging Device for Monitoring Mesenchymal Stromal Cells in Osteoarthritis Treatment
Brief Title: Handheld MPI Imaging to Track Stem Cells in Osteoarthritis
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soochow University (Other)
Responsible Party: Principal Investigator, Tuo Shao, Professor, Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KXXSC2025-IIT-23
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Knee Arthritis Osteoarthritis
MeSH Terms: interventions — Ferrosoferric Oxide; ferric oxide; Solutions; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UC-MSCs + SPIO + MPI Monitoring Group (Experimental): Participants in this group will receive a single intra-articular injection of ferumoxytol (SPIO)-labeled human umbilical cord-derived mesenchymal stromal cells (UC-MSCs, "TriCellPr-AC07" injection, 5-6×10^7 cells). The injection will be guided in real-time by a handheld Magnetic Particle Imaging (MPI) device to ensure accurate placement. Participants will undergo longitudinal MPI scans (at Day 1, 3, 7, and 30 post-injection) to quantitatively monitor the distribution, retention, and signal decay (as a surrogate for cell survival) of the labeled cells. Standard MRI will also be performed at baseline and follow-up to assess structural changes in cartilage and synovium. Clinical outcomes (WOMAC, VAS, SF-36) will be assessed by blinded evaluators.
  Interventions: Biological: Human Umbilical Cord-derived Mesenchymal Stromal Cells (hUC-MSCs)
- Placebo (SPIO Solution) Control Group (Placebo Comparator): Participants in this control group will receive a single intra-articular injection of an equivalent volume of ferumoxytol (SPIO) solution without mesenchymal stromal cells. The injection procedure, including the use of the handheld MPI device for real-time guidance, will be identical to the experimental group to maintain blinding. Participants will undergo the same schedule of MPI and MRI scans as the experimental group, as well as identical clinical assessments by blinded evaluators. This group serves to control for the potential effects of the injection procedure and the SPIO tracer itself.
  Interventions: Other: Ferumoxytol (SPIO) Solution for Injection (Placebo)

INTERVENTIONS:
Biological: Human Umbilical Cord-derived Mesenchymal Stromal Cells (hUC-MSCs) — This clinical trial evaluates an integrated cell therapy and imaging protocol for knee osteoarthritis. The core intervention is a single intra-articular injection of ferumoxytol (SPIO)-labeled human umbilical cord-derived mesenchymal stromal cells (MSCs), administered under real-time image guidance using a handheld Magnetic Particle Imaging (MPI) scanner. Its unique features are: 1) Real-time MPI-guided delivery for precise joint cavity targeting; 2) Subsequent use of the same MPI technology for serial quantitative monitoring of cell distribution, retention, and signal decay in vivo; 3) Use of the clinically approved agent ferumoxytol as an MPI tracer. This theragnostic approach combines therapeutic cells with a matched imaging modality for guided delivery and longitudinal tracking, distinguishing it from standard blind injections or studies using MRI only for anatomical assessment.
  Arms: UC-MSCs + SPIO + MPI Monitoring Group
Other: Ferumoxytol (SPIO) Solution for Injection (Placebo) — Single intra-articular injection of ferumoxytol (superparamagnetic iron oxide, SPIO) solution, without mesenchymal stromal cells. This serves as the placebo control. The injection is performed under real-time image guidance using the same handheld Magnetic Particle Imaging (MPI) scanner as the experimental group, and participants undergo identical MPI and MRI scanning schedules.
  Arms: Placebo (SPIO Solution) Control Group

SUMMARY:
This clinical trial aims to evaluate the use of a handheld Magnetic Particle Imaging (MPI) device for real-time, non-invasive monitoring of human umbilical cord-derived mesenchymal stromal cells (UC-MSCs) in patients with knee osteoarthritis (OA). The primary objective is to visualize and quantify the distribution, retention, and survival of SPIO (superparamagnetic iron oxide)-labeled MSCs within the joint space following intra-articular injection. By correlating MPI signal dynamics with established clinical outcomes (e.g., WOMAC, VAS scores) and anatomical MRI assessments, the study seeks to predict treatment efficacy and optimize therapeutic strategies for OA.

Current assessment of MSC therapy relies largely on MRI for structural evaluation, which has limited sensitivity for tracking early cell viability and migration. MPI offers high-contrast, radiation-free functional imaging capable of directly detecting SPIO-labeled cells. This study will enroll patients with mild-to-moderate OA (Kellgren-Lawrence grade II-III). Participants will receive a single injection of ferumoxytol-labeled UC-MSCs into the affected knee. MPI scans will be performed at multiple timepoints (day 1, 3, 7, and 30) to monitor cell homing, retention rate, and signal decay. MRI will be used in parallel to evaluate cartilage morphology and synovial changes.

The study expects to demonstrate that MPI can effectively track MSC behavior in vivo, providing a novel tool to understand cell therapy mechanisms, assess treatment response early, and potentially guide personalized OA management.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of knee osteoarthritis according to internationally accepted criteria (e.g., American College of Rheumatology criteria).
2. Age between 18 and 75 years, inclusive.
3. Radiographic Kellgren-Lawrence grade II or III in the target knee.
4. Chronic knee pain of arthritic origin.
5. Absence of local or systemic infection.
6. No contraindications to joint cavity puncture as determined by hematological and biochemical tests.
7. Willing and able to understand the study, provide informed consent, and comply with all study procedures.

Exclusion Criteria:

1. Lack of legal capacity or impaired capacity to provide informed consent.
2. Known active infection with HIV, hepatitis B virus, hepatitis C virus, or syphilis (positive serology).
3. Body mass index (BMI) > 30 kg/m².
4. Congenital or acquired deformity of the target knee.
5. Pregnant or breastfeeding women.
6. History of or current active malignancy.
7. Known immunodeficiency disorder.
8. Intra-articular injection (e.g., corticosteroids, hyaluronic acid) in the target knee within the past 3 months.
9. Concurrent participation in another interventional clinical trial.
10. Any other condition that, in the opinion of the investigator, would make the participant unsuitable for the study (e.g., significant comorbid illness).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
MPI-Based Joint Cavity Retention Rate of SPIO-labeled hUC-MSCs | Baseline (pre-injection) to Day 7 post-injection
  The percentage of the total injected Magnetic Particle Imaging (MPI) signal that remains within the target knee joint cavity at Day 7 post-injection. This quantitative measure, calculated using specialized MPI analysis software (e.g., Magnetic Particle Imaging Lab toolbox), serves as a primary indicator of successful cell homing and initial localization at the intended therapeutic site.

SECONDARY OUTCOMES:
Change in WOMAC Total Score | Baseline to Week 6 post-injection
  Change from baseline in the total score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC is a validated patient-reported outcome measure assessing pain (5 items), stiffness (2 items), and physical function (17 items) in knee osteoarthritis. Scores range from 0 (best) to 96 (worst). A negative change indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Tuo Shao, Study Director — Soochow University
Locations (1):
- Hainan General Hospital, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the primary publication of this study will be made available. This will include clinical outcomes (e.g., WOMAC, VAS scores), MRI assessment data, and quantitative MPI-derived metrics (e.g., signal retention rate, decay rate).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 3 months after main results publication. Ending 36 months after publication.
Access Criteria: Data access requests should be directed to the corresponding author or the designated data custodian at Hainan Provincial People's Hospital. Requestors will need to submit a methodologically sound research proposal for review by the study's Steering Committee. Access will be granted upon approval of the proposal and execution of a Data Use/Transfer Agreement.

REFERENCES:
- [Background] Feng X, Gao P, Li Y, Hui H, Jiang J, Xie F, Tian J. First magnetic particle imaging to assess pulmonary vascular leakage in vivo in the acutely injured and fibrotic lung. Bioeng Transl Med. 2023 Nov 29;9(2):e10626. doi: 10.1002/btm2.10626. eCollection 2024 Mar. PMID 38435827
- [Background] Ferreira-Filho VC, Morais B, Vieira BJC, Waerenborgh JC, Carmezim MJ, Toth CN, Meme S, Lacerda S, Jaque D, Sousa CT, Campello MPC, Pereira LCJ. Influence of SPION Surface Coating on Magnetic Properties and Theranostic Profile. Molecules. 2024 Apr 17;29(8):1824. doi: 10.3390/molecules29081824. PMID 38675647
- [Background] Nejadnik H, Tseng J, Daldrup-Link H. Magnetic resonance imaging of stem cell-macrophage interactions with ferumoxytol and ferumoxytol-derived nanoparticles. Wiley Interdiscip Rev Nanomed Nanobiotechnol. 2019 Jul;11(4):e1552. doi: 10.1002/wnan.1552. Epub 2019 Feb 7. PMID 30734542
- [Background] Matas J, Garcia C, Poblete D, Vernal R, Ortloff A, Luque-Campos N, Hidalgo Y, Cuenca J, Infante C, Cadiz MI, Khoury M, Luz-Crawford P, Espinoza F. A Phase I Dose-Escalation Clinical Trial to Assess the Safety and Efficacy of Umbilical Cord-Derived Mesenchymal Stromal Cells in Knee Osteoarthritis. Stem Cells Transl Med. 2024 Mar 15;13(3):193-203. doi: 10.1093/stcltm/szad088. PMID 38366909
- [Background] Pico OA, Espinoza F, Cadiz MI, Sossa CL, Becerra-Bayona SM, Salgado MCC, Rodriguez JER, Cardenas OFV, Cure JMQ, Khoury M, Arango-Rodriguez ML. Efficacy of a single dose of cryopreserved human umbilical cord mesenchymal stromal cells for the treatment of knee osteoarthritis:a randomized, controlled, double-blind pilot study. Cytotherapy. 2025 Feb;27(2):188-200. doi: 10.1016/j.jcyt.2024.09.005. Epub 2024 Oct 16. PMID 39503681
- [Background] Negoro T, Takagaki Y, Okura H, Matsuyama A. Trends in clinical trials for articular cartilage repair by cell therapy. NPJ Regen Med. 2018 Oct 11;3:17. doi: 10.1038/s41536-018-0055-2. eCollection 2018. PMID 30345076
- [Background] Xiang XN, Zhu SY, He HC, Yu X, Xu Y, He CQ. Mesenchymal stromal cell-based therapy for cartilage regeneration in knee osteoarthritis. Stem Cell Res Ther. 2022 Jan 10;13(1):14. doi: 10.1186/s13287-021-02689-9. PMID 35012666
- [Background] Vina ER, Kwoh CK. Epidemiology of osteoarthritis: literature update. Curr Opin Rheumatol. 2018 Mar;30(2):160-167. doi: 10.1097/BOR.0000000000000479. PMID 29227353
- [Background] Scheuing WJ, Reginato AM, Deeb M, Acer Kasman S. The burden of osteoarthritis: Is it a rising problem? Best Pract Res Clin Rheumatol. 2023 Jun;37(2):101836. doi: 10.1016/j.berh.2023.101836. Epub 2023 Aug 24. PMID 37633827
- [Background] Allen KD, Thoma LM, Golightly YM. Epidemiology of osteoarthritis. Osteoarthritis Cartilage. 2022 Feb;30(2):184-195. doi: 10.1016/j.joca.2021.04.020. Epub 2021 Sep 14. PMID 34534661